CLINICAL TRIAL: NCT00945152
Title: Topical MRSA Bactericidal Gel to Eliminate MRSA and Promote Accelerated Healing of cSSTI of Open Wounds
Brief Title: Effects of MRSA Bactericidal Gel To Promote Healing and Eliminate MRSA in cSSTI Vancogel(TM)
Acronym: Vancogel(R)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert S Berman MD (Other)
Responsible Party: Sponsor-Investigator, Robert S Berman MD, Sponsor-Investigator, Robert S Berman MD
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WIRB study # 1111446; None yet, self funding
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Bacterial Infections; Wounds
Keywords: Elimination of MRSA in open wounds; MRSA infected open wounds
MeSH Terms: conditions — Bacterial Infections; Wounds and Injuries | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Vancogel,Treatment,Kill MRSA,Heal (Experimental): Treatment of open wounds with Vancogel(R) 1.25-1.50% to eliminate MRSA. End point is: a negative culture report after 1-3 topical applications. The infected wounds with MRSA will be treated with the Vancomycin 1.25 to 1.50% complex gel formulation and will have conventional management in order to heal the wound. Vancogel is anticipated to accelerate wound healing by eliminating MRSA. A randomized, double blind study protocol approved by FDA.
  Interventions: Drug: Vancomycin 1.25-1.50% in a complex gel formulation trademarked Vancogel(R)
- Placebo (Placebo Comparator): Half of the patients in the study will be given a placebo consisting of all ingredients in Vancogel except the active principal Vancomycin in order to compare their clinical efficacy in rate of wound healingafter 1-3 applications
  Interventions: Drug: Placebo, complex gel formulation without Vancomycin

INTERVENTIONS:
Drug: Vancomycin 1.25-1.50% in a complex gel formulation trademarked Vancogel(R) — Topical use for open wounds culturing out MRSA. One to three applications of the compound over a weeks time. Consists of Vancomycin 1.25-1.50% in a complex gel formulation.
  Other Names: Vancogel (R)# 77708836/Trademark issued 12-11-2012 Patent issued 02-02-2016 # 9248159; Topical MRSA Bactericidal Gel; Vancomycin complex gel formulation
  Arms: Drug Vancogel,Treatment,Kill MRSA,Heal
Drug: Placebo, complex gel formulation without Vancomycin — Complex gel formulation applied as the placebo and is unknown because of the trial design. Complex gel formulation without Vancomycin
  Other Names: Safgel
  Arms: Placebo

SUMMARY:
Based on personal experience and the literature it is reasonable expectation that Vancomycin is a viable treatment in a direct contact form to eliminate MRSA from open wounds in order to heal the wounds by conventional means. The key question in my research has been to measure the effectiveness of my Vancomycin Gel by culturing the wound, applying the Gel in a controlled manner and then culturing the wound after one week. The end point to achieve in the process, is a clinical response of accelerated healing and negative culture report. Another question to solve is the duration of potency and stability of the Vancomycin gel over time.

DETAILED DESCRIPTION:
Over a prior preliminary 33 month study I have found negative cultures at the end of one week of treatment and have had microbiological studies establishing the same MIC zones in culture media greater than 15mm over a 33 month time frame. The microbiological and HPLC studies are completed at present and approved. I have started the phase 2 studies on August 1,2011 as authorized by the FDA on June 22,2011.

ELIGIBILITY:
Inclusion Criteria:

* MRSA infected open wounds
* Acute and chronic wounds
* Type of wounds: venous stasis,diabetic, pressure, post surgical, post traumatic, and spontaneous
* Infection criteria: Include a positive culture for MRSA
* Location of ulcers: any place on the body
* Diagnosis of MRSA: Based on tissue cultures of MRSA
* Willing and reliable patients
* Study to include only one ulceration no more than 50 square centimeters
* The study to include stages two and three ulcerations

Exclusion Criteria:

* Non-compliant patients
* Patient must accept all issues in consent form
* Non compliance to include failed appointments
* Wounds greater than 50sq. cm
* No wounds deeper than soft tissue
* Ischemic or vascular disease, dermatitis, immune deficiency,or psoriasis
* Allergy to Vancomycin
* Post irradiation ulceration
* Bleeding disorders
* Skin allergies to adhesives and tape
* Ulcers related to cancers
* Multiple wounds
* Stage 4 ulcerations
* Patients in any other trial
* Patients with any other conditions which, in the opinion of the investigator/doctor, would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Eliminate MRSA infection | One week
  Cultures taken during and prior to treatment and after.

SECONDARY OUTCOMES:
More rapid healing of cSSTI | 3 weeks
  The effects of the MRSA bactericidal gel will accelerate wound healing by eliminating the infection in cSSTI wounds

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Berman, MD, Principal Investigator
Locations (1):
- Robert S Berman MD /661 Maplewood Drive #21, Jupiter, Florida, United States